CLINICAL TRIAL: NCT01902381
Title: A Pilot Study of CPI-613 in Patients With Myelodysplastic Syndrome Who Have Failed Previous Therapy
Brief Title: CPI-613 in Treating Patients With Myelodysplastic Syndromes Who Failed Previous Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug sponsor suspended study prematurely then study was terminated. Expected enrollment was not met.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00024007; NCI-2013-01312 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA012197 (NIH); CCCWFU 29113 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Previously Treated Myelodysplastic Syndromes
MeSH Terms: interventions — devimistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (6, 8-bis(benzylthio) octanoic acid) (Experimental): Patients receive treatment 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1 and 4 of weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 6,8-bis(benzylthio)octanoic acid

INTERVENTIONS:
Drug: 6,8-bis(benzylthio)octanoic acid — Given IV
  Other Names: alpha-lipoic acid analogue CPI-613; CPI-613

SUMMARY:
This pilot clinical trial studies 6, 8-bis (benzylthio) octanoic acid (CPI-613) in treating patients with myelodysplastic syndromes who failed previous therapy. Sometimes when chemotherapy or biological therapy is given, it does not stop the growth of tumor cells. The tumor is said to be resistant to treatment. 6, 8-bis (benzylthio) octanoic acid may interfere with the growth of tumor cells and may be an effective treatment for myelodysplastic syndromes that did not respond to previous therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and anti-cancer activities of CPI-613 in myelodysplastic syndrome (MDS) patients who have failed previous agents (such as decitabine [Dacogen], azacitidine [Vidaza], growth factors or lenalidomide).

OUTLINE:

Patients receive 6, 8-bis (benzylthio) octanoic acid intravenously (IV) over 2 hours on days 1 and 4 of weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented MDS of any risk group that has failed previous therapy (therapy failure is defined as patients who have been sufficiently treated with previous agents without response in the opinion of the treating physician, or whose disease has progressed or relapsed while on a hypomethylating agent)
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 3
* Expected survival > 2 months
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists
* Patients must have fully recovered from the acute, non-hematological, non-infectious toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities; patients with persisting, non-hematologic, non-infectious toxicities from prior treatment =< grade 2 are eligible, but must be documented as such
* Aspartate aminotransferase (AST/serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x upper normal limit (UNL)
* Alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 3 x UNL (=< 5x ULN if liver metastases present)
* Bilirubin =< 1.5 x UNL
* Serum creatinine =< 1.5 mg/dL or 133 umol/L
* International normalized ratio (or INR) must be < 1.5
* Albumin >= 2.0 g/dL or >= 20 g/L
* Mentally competent, ability to understand and willingness to sign an Institutional Review Board (IRB)-approved written informed consent form
* Have access via central line (e.g., portacath)

Exclusion Criteria:

* Serious medical illness, such as significant cardiac disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, coronary artery disease, myocardial infarction within the past 3 months, uncontrolled cardiac arrhythmia, pericardial disease or New York Heart Association class III or IV), or severe debilitating pulmonary disease, that would potentially increase patients' risk for toxicity
* Patients with active central nervous system (CNS) or epidural tumor
* Any active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease)
* Any condition or abnormality which may, in the opinion of the investigator, compromise his or her safety
* Pregnant women, or women of child-bearing potential not using reliable means of contraception
* Fertile men unwilling to practice contraceptive methods during the study period
* Lactating females
* Life expectancy less than 2 months
* Unwilling or unable to follow protocol requirements
* A history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome, etc.)
* Evidence of active infection or serious infection within the past month
* Requirement for immediate palliative treatment of any kind including surgery
* Prior illicit drug addiction
* Patients with large and recurrent pleural or peritoneal effusions requiring frequent drainage (e.g. weekly)
* Patients with any amount of clinically significant pericardial effusion
* Patients with known human immunodeficiency virus (HIV) infection; (Note: patients with known HIV infection are excluded because patients with an immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, and because there may be unknown or dangerous drug interactions between CPI-613 and anti-retroviral agents used to treat HIV infections)
* Patients who have received radiotherapy, surgery, treatment with cytotoxic agents (except CPI-613), treatment with biologic agents, immunotherapy, or any other anti-cancer therapy of any kind, or any other standard or investigational treatment for their cancer, or any other investigational agent for any indication, within the past 2 weeks prior to initiation of CPI-613 treatment
* Patients that have received a chemotherapy regimen with stem cell support in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pardee, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (6, 8-bis(Benzylthio) Octanoic Acid)
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (6, 8-bis(Benzylthio) Octanoic Acid)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR), Defined as the Combined Rate of Complete Remission (CR), Marrow CR, Partial Remission (PR), or Stable Disease (SD), as Described by Cheson, et al. (2006)
Description: Response rate (RR), defined as the combined of complete remission (CR), marrow CR, partial remission (PR), or stable disease (SD), as described by Cheson, et al. (2006). The number of patients achieving RR will be presented.
  Complete remission - Bone marrow: ≤ 5% myeloblasts with normal maturation of all cell lines; Marrow CR - Bone marrow: ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment Partial remission - All CR criteria if abnormal before treatment except: Bone marrow blasts decreased by ≥ 50% over pretreatment but still > 5%, cellularity and morphology not relevant Stable disease - Failure to achieve at least PR, but no evidence of progression for > 8 wks
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (6, 8-bis(Benzylthio) Octanoic Acid)
Number analyzed (Participants) | 12
Participants | 11

2. Secondary Outcome: Safety Profile of CPI-613, Based on Evaluation of Symptoms, Vital Signs, ECOG Performance Status and Survival, Clinical Chemistry, Hematology, and Coagulation, Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events v 4.0
Description: Safety profile of CPI-613, based on evaluation of symptoms, vital signs, ECOG performance status and survival, clinical chemistry, hematology, and coagulation, assessed by National Cancer Institute Common Terminology Criteria for Adverse Events v 4.0. Toxicities related to the treatment will be examined by looking at each toxicity identified by grade (highest grade of each toxicity per patient so that there is only one event attributed to each patient for a given toxicity).
Time Frame: During treatment, a median of 4 months with a maximum of 40 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (6, 8-bis(Benzylthio) Octanoic Acid)
Number analyzed (Participants) | 12
Participants
  Anemia: Unobserved | 5
  Anemia: Grade 1 | 0
  Anemia: Grade 2 | 2
  Anemia: Grade 3 | 2
  Anemia: Grade 4 | 3
  Febrile neutropenia: Unobserved | 11
  Febrile neutropenia: Grade 1 | 0
  Febrile neutropenia: Grade 2 | 0
  Febrile neutropenia: Grade 3 | 1
  Febrile neutropenia: Grade 4 | 0
  Sinus bradycardia: Unobserved | 11
  Sinus bradycardia: Grade 1 | 0
  Sinus bradycardia: Grade 2 | 0
  Sinus bradycardia: Grade 3 | 1
  Sinus bradycardia: Grade 4 | 0
  Cardiac disorders - Other: Unobserved | 11
  Cardiac disorders - Other: Grade 1 | 0
  Cardiac disorders - Other: Grade 2 | 0
  Cardiac disorders - Other: Grade 3 | 0
  Cardiac disorders - Other: Grade 4 | 1
  Dry eye: Unobserved | 11
  Dry eye: Grade 1 | 1
  Dry eye: Grade 2 | 0
  Dry eye: Grade 3 | 0
  Dry eye: Grade 4 | 0
  Eye disorders - Other: Unobserved | 11
  Eye disorders - Other: Grade 1 | 1
  Eye disorders - Other: Grade 2 | 0
  Eye disorders - Other: Grade 3 | 0
  Eye disorders - Other: Grade 4 | 0
  Eye disorders - Right eye subconjunctival hemorrhage: Unobserved | 11
  Eye disorders - Right eye subconjunctival hemorrhage: Grade 1 | 1
  Eye disorders - Right eye subconjunctival hemorrhage: Grade 2 | 0
  Eye disorders - Right eye subconjunctival hemorrhage: Grade 3 | 0
  Eye disorders - Right eye subconjunctival hemorrhage: Grade 4 | 0
  Constipation: Unobserved | 10
  Constipation: Grade 1 | 2
  Constipation: Grade 2 | 0
  Constipation: Grade 3 | 0
  Constipation: Grade 4 | 0
  Diarrhea: Unobserved | 1
  Diarrhea: Grade 1 | 5
  Diarrhea: Grade 2 | 5
  Diarrhea: Grade 3 | 1
  Diarrhea: Grade 4 | 0
  Gastroesophageal reflux disease: Unobserved | 11
  Gastroesophageal reflux disease: Grade 1 | 1
  Gastroesophageal reflux disease: Grade 2 | 0
  Gastroesophageal reflux disease: Grade 3 | 0
  Gastroesophageal reflux disease: Grade 4 | 0
  Nausea: Unobserved | 4
  Nausea: Grade 1 | 5
  Nausea: Grade 2 | 3
  Nausea: Grade 3 | 0
  Nausea: Grade 4 | 0
  Taste alteration (dysgeusia): Unobserved | 11
  Taste alteration (dysgeusia): Grade 1 | 1
  Taste alteration (dysgeusia): Grade 2 | 0
  Taste alteration (dysgeusia): Grade 3 | 0
  Taste alteration (dysgeusia): Grade 4 | 0
  Vomiting: Unobserved | 8
  Vomiting: Grade 1 | 4
  Vomiting: Grade 2 | 0
  Vomiting: Grade 3 | 0
  Vomiting: Grade 4 | 0
  Chills: Unobserved | 11
  Chills: Grade 1 | 1
  Chills: Grade 2 | 0
  Chills: Grade 3 | 0
  Chills: Grade 4 | 0
  Edema limbs: Unobserved | 10
  Edema limbs: Grade 1 | 2
  Edema limbs: Grade 2 | 0
  Edema limbs: Grade 3 | 0
  Edema limbs: Grade 4 | 0
  Fatigue: Unobserved | 5
  Fatigue: Grade 1 | 2
  Fatigue: Grade 2 | 3
  Fatigue: Grade 3 | 2
  Fatigue: Grade 4 | 0
  Fever: Unobserved | 9
  Fever: Grade 1 | 3
  Fever: Grade 2 | 0
  Fever: Grade 3 | 0
  Fever: Grade 4 | 0
  Malaise: Unobserved | 11
  Malaise: Grade 1 | 1
  Malaise: Grade 2 | 0
  Malaise: Grade 3 | 0
  Malaise: Grade 4 | 0
  Lung infection: Unobserved | 11
  Lung infection: Grade 1 | 0
  Lung infection: Grade 2 | 0
  Lung infection: Grade 3 | 1
  Lung infection: Grade 4 | 0
  Mucosal infection: Unobserved | 11
  Mucosal infection: Grade 1 | 1
  Mucosal infection: Grade 2 | 0
  Mucosal infection: Grade 3 | 0
  Mucosal infection: Grade 4 | 0
  Sinusitis: Unobserved | 11
  Sinusitis: Grade 1 | 0
  Sinusitis: Grade 2 | 1
  Sinusitis: Grade 3 | 0
  Sinusitis: Grade 4 | 0
  Bruising: Unobserved | 11
  Bruising: Grade 1 | 1
  Bruising: Grade 2 | 0
  Bruising: Grade 3 | 0
  Bruising: Grade 4 | 0
  Alanine aminotransferase increased: Unobserved | 9
  Alanine aminotransferase increased: Grade 1 | 3
  Alanine aminotransferase increased: Grade 2 | 0
  Alanine aminotransferase increased: Grade 3 | 0
  Alanine aminotransferase increased: Grade 4 | 0
  Alkaline phosphatase increased: Unobserved | 10
  Alkaline phosphatase increased: Grade 1 | 2
  Alkaline phosphatase increased: Grade 2 | 0
  Alkaline phosphatase increased: Grade 3 | 0
  Alkaline phosphatase increased: Grade 4 | 0
  Aspartate aminotransferase increased: Unobserved | 9
  Aspartate aminotransferase increased: Grade 1 | 3
  Aspartate aminotransferase increased: Grade 2 | 0
  Aspartate aminotransferase increased: Grade 3 | 0
  Aspartate aminotransferase increased: Grade 4 | 0
  Blood bilirubin increased: Unobserved | 11
  Blood bilirubin increased: Grade 1 | 1
  Blood bilirubin increased: Grade 2 | 0
  Blood bilirubin increased: Grade 3 | 0
  Blood bilirubin increased: Grade 4 | 0
  Creatinine increased: Unobserved | 11
  Creatinine increased: Grade 1 | 0
  Creatinine increased: Grade 2 | 0
  Creatinine increased: Grade 3 | 1
  Creatinine increased: Grade 4 | 0
  Electrocardiogram QT corrected interval prolonged: Unobserved | 11
  Electrocardiogram QT corrected interval prolonged: Grade 1 | 1
  Electrocardiogram QT corrected interval prolonged: Grade 2 | 0
  Electrocardiogram QT corrected interval prolonged: Grade 3 | 0
  Electrocardiogram QT corrected interval prolonged: Grade 4 | 0
  Lymphocyte count decreased: Unobserved | 7
  Lymphocyte count decreased: Grade 1 | 1
  Lymphocyte count decreased: Grade 2 | 1
  Lymphocyte count decreased: Grade 3 | 2
  Lymphocyte count decreased: Grade 4 | 1
  Lymphocyte count increased: Unobserved | 11
  Lymphocyte count increased: Grade 1 | 0
  Lymphocyte count increased: Grade 2 | 0
  Lymphocyte count increased: Grade 3 | 1
  Lymphocyte count increased: Grade 4 | 0
  Neutrophil count decreased: Unobserved | 7
  Neutrophil count decreased: Grade 1 | 0
  Neutrophil count decreased: Grade 2 | 0
  Neutrophil count decreased: Grade 3 | 1
  Neutrophil count decreased: Grade 4 | 4
  Platelet count decreased: Unobserved | 6
  Platelet count decreased: Grade 1 | 0
  Platelet count decreased: Grade 2 | 1
  Platelet count decreased: Grade 3 | 1
  Platelet count decreased: Grade 4 | 4
  White blood cell decreased: Unobserved | 6
  White blood cell decreased: Grade 1 | 0
  White blood cell decreased: Grade 2 | 2
  White blood cell decreased: Grade 3 | 3
  White blood cell decreased: Grade 4 | 1
  Anorexia: Unobserved | 9
  Anorexia: Grade 1 | 0
  Anorexia: Grade 2 | 3
  Anorexia: Grade 3 | 0
  Anorexia: Grade 4 | 0
  Hypercalcemia: Unobserved | 11
  Hypercalcemia: Grade 1 | 1
  Hypercalcemia: Grade 2 | 0
  Hypercalcemia: Grade 3 | 0
  Hypercalcemia: Grade 4 | 0
  Hyperglycemia: Unobserved | 8
  Hyperglycemia: Grade 1 | 2
  Hyperglycemia: Grade 2 | 1
  Hyperglycemia: Grade 3 | 1
  Hyperglycemia: Grade 4 | 0
  Hypoalbuminemia: Unobserved | 10
  Hypoalbuminemia: Grade 1 | 0
  Hypoalbuminemia: Grade 2 | 2
  Hypoalbuminemia: Grade 3 | 0
  Hypoalbuminemia: Grade 4 | 0
  Hypocalcemia: Unobserved | 11
  Hypocalcemia: Grade 1 | 0
  Hypocalcemia: Grade 2 | 1
  Hypocalcemia: Grade 3 | 0
  Hypocalcemia: Grade 4 | 0
  Hypomagnesemia: Unobserved | 9
  Hypomagnesemia: Grade 1 | 3
  Hypomagnesemia: Grade 2 | 0
  Hypomagnesemia: Grade 3 | 0
  Hypomagnesemia: Grade 4 | 0
  Hyponatremia: Unobserved | 10
  Hyponatremia: Grade 1 | 2
  Hyponatremia: Grade 2 | 0
  Hyponatremia: Grade 3 | 0
  Hyponatremia: Grade 4 | 0
  Generalized muscle weakness: Unobserved | 8
  Generalized muscle weakness: Grade 1 | 0
  Generalized muscle weakness: Grade 2 | 2
  Generalized muscle weakness: Grade 3 | 2
  Generalized muscle weakness: Grade 4 | 0
  Pain in extremity: Unobserved | 11
  Pain in extremity: Grade 1 | 0
  Pain in extremity: Grade 2 | 1
  Pain in extremity: Grade 3 | 0
  Pain in extremity: Grade 4 | 0
  Musculoskeletal and connective tissue disorder - Other: Unobserved | 11
  Musculoskeletal and connective tissue disorder - Other: Grade 1 | 0
  Musculoskeletal and connective tissue disorder - Other: Grade 2 | 1
  Musculoskeletal and connective tissue disorder - Other: Grade 3 | 0
  Musculoskeletal and connective tissue disorder - Other: Grade 4 | 0
  Cognitive disturbance: Unobserved | 11
  Cognitive disturbance: Grade 1 | 1
  Cognitive disturbance: Grade 2 | 0
  Cognitive disturbance: Grade 3 | 0
  Cognitive disturbance: Grade 4 | 0
  Dizziness: Unobserved | 11
  Dizziness: Grade 1 | 1
  Dizziness: Grade 2 | 0
  Dizziness: Grade 3 | 0
  Dizziness: Grade 4 | 0
  Dysgeusia: Unobserved | 11
  Dysgeusia: Grade 1 | 1
  Dysgeusia: Grade 2 | 0
  Dysgeusia: Grade 3 | 0
  Dysgeusia: Grade 4 | 0
  Lethargy: Unobserved | 11
  Lethargy: Grade 1 | 0
  Lethargy: Grade 2 | 1
  Lethargy: Grade 3 | 0
  Lethargy: Grade 4 | 0
  Memory impairment: Unobserved | 11
  Memory impairment: Grade 1 | 1
  Memory impairment: Grade 2 | 0
  Memory impairment: Grade 3 | 0
  Memory impairment: Grade 4 | 0
  Seizure: Unobserved | 11
  Seizure: Grade 1 | 0
  Seizure: Grade 2 | 1
  Seizure: Grade 3 | 0
  Seizure: Grade 4 | 0
  Hematuria: Unobserved | 11
  Hematuria: Grade 1 | 0
  Hematuria: Grade 2 | 1
  Hematuria: Grade 3 | 0
  Hematuria: Grade 4 | 0
  Renal and urinary disorders - Other: Unobserved | 11
  Renal and urinary disorders - Other: Grade 1 | 0
  Renal and urinary disorders - Other: Grade 2 | 0
  Renal and urinary disorders - Other: Grade 3 | 1
  Renal and urinary disorders - Other: Grade 4 | 0
  Dyspnea: Unobserved | 10
  Dyspnea: Grade 1 | 0
  Dyspnea: Grade 2 | 1
  Dyspnea: Grade 3 | 1
  Dyspnea: Grade 4 | 0
  Epistaxis: Unobserved | 11
  Epistaxis: Grade 1 | 1
  Epistaxis: Grade 2 | 0
  Epistaxis: Grade 3 | 0
  Epistaxis: Grade 4 | 0
  Erythema multiforme: Unobserved | 11
  Erythema multiforme: Grade 1 | 0
  Erythema multiforme: Grade 2 | 1
  Erythema multiforme: Grade 3 | 0
  Erythema multiforme: Grade 4 | 0
  Skin and subcutaneous tissue disorders - Dry Skin: Unobserved | 11
  Skin and subcutaneous tissue disorders - Dry Skin: Grade 1 | 1
  Skin and subcutaneous tissue disorders - Dry Skin: Grade 2 | 0
  Skin and subcutaneous tissue disorders - Dry Skin: Grade 3 | 0
  Skin and subcutaneous tissue disorders - Dry Skin: Grade 4 | 0
  Hypotension: Unobserved | 10
  Hypotension: Grade 1 | 1
  Hypotension: Grade 2 | 0
  Hypotension: Grade 3 | 1
  Hypotension: Grade 4 | 0

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Survival curves for PFS using Kaplan-Meier techniques will be estimated. In addition, the 6 month and 1-year PFS rates for these participants will be estimated.
  Disease progression: For patients with:
  Less than 5% blasts: ≥ 50% increase in blasts to > 5% blasts 5%-10% blasts: ≥ 50% increase to > 10% blasts 10%-20% blasts: ≥ 50% increase to > 20% blasts 20%-30% blasts: ≥ 50% increase to > 30% blasts
  Any of the following:
  At least 50% decrement from maximum remission/response in granulocytes or platelets Reduction in Hgb by ≥ 2 g/dL Transfusion dependence
  Survival Endpoints:
  Overall: death from any cause Event free: failure or death from any cause PFS: disease progression or death from MDS DFS: time to relapse Cause-specific death: death related to MDS
Time Frame: 6 and 12 months post treatment start
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment (6, 8-bis(Benzylthio) Octanoic Acid)
Number analyzed (Participants) | 12
Percentage of participants
  6 Month | 65.6 [38.2 to 93.1]
  12 Month | 46.9 [17.4 to 76.3]

4. Secondary Outcome: Overall Survival (OS)
Description: Survival curves for OS using Kaplan-Meier techniques will be estimated. In addition, the 6 month and 1-year OS rates for these participants will be estimated.
Time Frame: 6 and 12 months post treatment start
Measure: Number (95% Confidence Interval); unit: overall survival percentage
Arm/Group | Treatment (6, 8-bis(Benzylthio) Octanoic Acid)
Number analyzed (Participants) | 12
overall survival percentage
  6 Month OS | 81.8 [59.0 to 100]
  12 Month OS | 54.6 [25.1 to 84.0]

5. Secondary Outcome: Number of Patients Who Achieve a Reduction in Blood Transfusion Requirements
Description: Number of patients who achieve a reduction in blood transfusion requirements.
Time Frame: Up to 5 years
Population: Patients with blood transfusions at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (6, 8-bis(Benzylthio) Octanoic Acid)
Number analyzed (Participants) | 9
Participants | 1

6. Secondary Outcome: Number of Patients Who Achieve Hematologic Improvement (HI), as Defined by Cheson, et al. (2006)
Description: Number of patients who achieve hematologic improvement (HI), as defined by Cheson, et al. (2006).
  Criteria:
  Erythroid response (pretreatment, < 11 g/dL) - Hgb increase by ≥ 1.5 g/dL.
  Platelet response (pretreatment, < 100 × 109/L) - Absolute increase of ≥ 30 × 109/L for patients starting with > 20 × 109/L platelets. Increase from < 20 × 109/L to > 20 × 109/L and by at least 100%
  Neutrophil response (pretreatment, < 1.0 × 109/L) - At least 100% increase and an absolute increase > 0.5 × 109/L
  Progression or relapse after HI - At least 1 of the following:
  At least 50% decrement from maximum response levels in granulocytes or platelets Reduction in Hgb by ≥ 1.5 g/dL
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (6, 8-bis(Benzylthio) Octanoic Acid)
Number analyzed (Participants) | 12
Participants | 3

ADVERSE EVENTS:
Time Frame: During treatment, a median of 4 months with a maximum of 40 months.
Description: Serious Adverse Events are defined as unexpected grade 4 and all grade 5
Arm/Group | Treatment (6, 8-bis(Benzylthio) Octanoic Acid)
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (6, 8-bis(Benzylthio) Octanoic Acid) (N=12)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Cardiac disorders - Other: (Cardiac disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (6, 8-bis(Benzylthio) Octanoic Acid) (N=12)
Anemia (Blood and lymphatic system disorders) | 12 (97)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (3)
Lymphopenia (1-5.1) (Blood and lymphatic system disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (3)
Cardiac disorders - Other: Murmur (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 4 (5)
Dry eye (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Eye disorders - Other: (Eye disorders) | 1 (1)
Eye disorders - Other: Right eye subconjunctival hemorrhage (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (7)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (23)
Diarrhea (Gastrointestinal disorders) | 12 (49)
Dry mouth (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 8 (27)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (2)
Rectal pain (Gastrointestinal disorders) | 2 (4)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5)
Gastrointestinal disorders - Other: (Gastrointestinal disorders) | 2 (4)
Gastrointestinal disorders - Other: Indigestion (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 3 (3)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 6 (12)
Fatigue (General disorders) | 11 (53)
Fever (General disorders) | 4 (6)
Gait disturbance (General disorders) | 4 (10)
Malaise (General disorders) | 4 (4)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 5 (7)
General disorders and administration site conditions - Other: (General disorders) | 2 (3)
General disorders and administration site conditions - Other: AE logs rec'd 2/18/15 (General disorders) | 1 (1)
Hepatobiliary disorders - Other: Hepatomegaly (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Immune system disorders - Other: (Immune system disorders) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 4 (5)
Mucosal infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (3)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (5)
Vaginal infection (Infections and infestations) | 1 (1)
Infections and infestations - Other: (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 5 (11)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Injury, poisoning and procedural complications - Other: (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 6 (12)
Alanine aminotransferase increased (Investigations) | 6 (41)
Alkaline phosphatase increased (Investigations) | 5 (12)
Aspartate aminotransferase increased (Investigations) | 7 (35)
Blood bilirubin increased (Investigations) | 7 (14)
Creatinine increased (Investigations) | 1 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (2)
Haptoglobin decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 12 (76)
Lymphocyte count increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 11 (61)
Platelet count decreased (Investigations) | 12 (96)
White blood cell decreased (Investigations) | 12 (74)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (13)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (93)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (21)
Hypocalcemia (Metabolism and nutrition disorders) | 8 (20)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 5 (12)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (23)
Hyponatremia (Metabolism and nutrition disorders) | 9 (25)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Iron overload (Metabolism and nutrition disorders) | 4 (4)
Metabolism and nutrition disorders - Other: (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (15)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other: (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 3 (7)
Dizziness (Nervous system disorders) | 6 (13)
Dysgeusia (Nervous system disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 2 (3)
Memory impairment (Nervous system disorders) | 3 (5)
Paresthesia (Nervous system disorders) | 1 (4)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Seizure (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (10)
Confusion (Psychiatric disorders) | 2 (3)
Depression (Psychiatric disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 5 (15)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 4 (5)
Urinary frequency (Renal and urinary disorders) | 3 (4)
Urinary incontinence (Renal and urinary disorders) | 3 (9)
Renal and urinary disorders - Other: (Renal and urinary disorders) | 3 (4)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (36)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other: (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other: (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other: Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other: log rec'd 3/17/15 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other: log rec'd 3/17/15/ Arm Wound (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 2 (6)
Hypotension (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT01902381/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT01902381/ICF_001.pdf